CLINICAL TRIAL: NCT07073456
Title: Viscoelastic Coagulation Monitor as an Early Index of Sepsis in Patients Admitted With Infection at the Emergency Department: The VISION Project
Brief Title: Viscoelastic Coagulation for Early Sepsis Detection
Acronym: VISION
Status: Recruiting | Type: Observational
Sponsor: Hellenic Institute for the Study of Sepsis (Other)
Responsible Party: Principal Investigator, Evangelos Giamarellos-Bourboulis, Professor of Internal Medicine and Infectious Diseases, 4th Department of Internal Medicine, NKUA, President of the European Sepsis Alliance, President of the Hellenic Institute for the Study of Sepsis, President of the Hellenic Society for Chemotherapy, National and Kapodistrian University of Athens
Other Study IDs: 10th/09-10-2024
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2024-10

CONDITIONS: Infection; Sepsis
Keywords: blood coagulation; infection; sepsis; clot formation; Viscoelastic Coagulation Monitor; early sepsis detection
MeSH Terms: conditions — Infections; Sepsis; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with suspicion of infection, defined according to medical judgment
  Interventions: Diagnostic Test: Viscoelastic Coagulation Monitoring measurements

INTERVENTIONS:
Diagnostic Test: Viscoelastic Coagulation Monitoring measurements — Peripheral venous blood samples will be obtained for the assessment of the eight following parameters utilizing the VCM (Viscoelastic Coagulation Monitor) device: clot time, clot formation time, alpha angle, amplitude at 10 minutes, amplitude at 20 minutes, maximum clot formation, lysis index at 30 minutes, and lysis index at 45 minutes. These parameters will be measured at the Emergency Department and subsequently on a daily basis for three consecutive days, if the patient is hospitalised.

SUMMARY:
The goal of this observational study is to investigate whether selected variables of coagulation measured by Viscoelastic Coagulation Monitoring (VCM) can serve as early predictors of progression to sepsis in adult patients presenting to the emergency department (ED) with suspected infection. The main questions it aims to answer are: Can any of the eight VCM-derived coagulation parameters predict early progression into sepsis? Is there a specific VCM profile associated with higher sepsis risk at ED presentation? Participants presenting to the Emergency Department with signs of suspected infection will be asked to provide written informed consent, either personally or via a legal representative. Upon consent, they will be enrolled in the study. All participants will undergo at the Emergency Department blood sampling for VCM analysis, for complete blood count, routine biochemical tests and inflammatory markers (e.g., CRP and procalcitonin). In case of discharge, patients will be contacted by phone for three consecutive days to monitor the course of infection and assess survival status. In case of admission, blood for VCM analysis will be collected daily for three consecutive days. This is a single-center, prospective proof-of-concept study conducted at ATTIKON University General Hospital in collaboration with the 4th Department of Internal Medicine.

ELIGIBILITY:
Inclusion Criteria:

* Adults male or female (age 18 years or more)
* Suspicion of infection, defined according to medical judgment

Exclusion Criteria:

* Age less than 18 years
* Denial for consent
* Intake of any anti-coagulant medication the last one month
* Intake of any anti-platelet medication the last one month
* Intake of any biological disease modifying anti-rheumatic medication the last one month
* Medical history of inflammatory bowel disease or pulmonary hypertension
* Any medical history of hemophilia or congenital coagulation disorders
* Any known solid tumor or hematologic malignancy irrespective the stage and treatment
* Known infection by the hepatitis viruses B and C
* Known infection by the human immunodeficiency virus
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, presenting to the Emergency Department of the General Hospital of Attikon, who meet all inclusion criteria and who do not meet any exclusion criterion will be enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-11-25 (Estimated)

PRIMARY OUTCOMES:
Difference in any variable captured by VCM between patients who progress or not into sepsis the first 72 hours. | From enrollment to 72-hour follow-up period
  The study primary endpoint is the difference in any variable captured by VCM between patients who progress or not into sepsis the first 72 hours. VCM measurements of any visit can be used for this endpoint.

SECONDARY OUTCOMES:
Difference in any variable captured by VCM between patients who progress or not into any major embolic event the first 72 hours | From enrollment to 72-hour-follow up period
  Difference in any variable captured by VCM between patients who progress or not into any major embolic event the first 72 hours.
Correlation between the eight VCM variables and the coagulation variables. | From enrollment to 72-hour-follow-up period
  Assessment of the correlation between eight viscoelastic parameters measured using the VCM® device and standard laboratory coagulation markers.
  The VCM parameters include: Clot Time (CT), Clot Formation Time (CFT), Alpha Angle (α), Amplitude at 10 minutes (A10), Amplitude at 20 minutes (A20), Maximum Clot Firmness (MCF), Lysis Index at 30 minutes (LI30), Lysis Index at 45 minutes (LI45).
  These will be correlated with the following coagulation variables:
  Absolute platelet count, International Normalized Ratio (INR), Activated Partial Thromboplastin Time (aPTT), D-dimers, Fibrinogen concentration.
  INR, aPTT, fibrinogen, and D-dimers will be measured using the SIEMENS coagulation panel. Correlation analysis will be performed using Spearman's rank correlation coefficient.
Correlation between the eight VCM variables and the measured inflammatory mediators | From enrollment to 72-hour-follow up period
  Assessment of the correlation between eight viscoelastic parameters measured using the VCM® device and inflammatory markers. The VCM parameters include: Clot Time (CT), Clot Formation Time (CFT), Alpha Angle (α), Amplitude at 10 minutes (A10), Amplitude at 20 minutes (A20), Maximum Clot Firmness (MCF), Lysis Index at 30 minutes (LI30), Lysis Index at 45 minutes (LI45). These will be correlated with the following inflammatory variables: tissue factor, suPAR, IL-1β, IL-6, IL-8 and TNFα.Tissue factor, suPAR, IL-1β, IL-6, IL-8 and TNFα will be measured in stored plasma samples by an enzyme immunosorbent assay. Correlation analysis will be performed using Spearman's rank correlation coefficient.

CONTACTS AND LOCATIONS:
Locations (1):
- ED & 4th Department of Internal Medicine, "Attikon" University Hospital, National and Kapodistrian University of Athens, Medical School, Chaïdári, Attica, Greece